CLINICAL TRIAL: NCT00691314
Title: Safety and Efficacy of Stent Implantation in Symptomatic Extra- and Intracranial Artery Stenosis
Brief Title: Efficacy and Safety of Stent Implantation in Symptomatic Extra- and Intracranial Artery Stenosis
Acronym: ESSCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Liying Cui, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006BAI01A10-2
Record Dates: First submitted 2008-04-12; First posted 2008-06-05 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Stroke; Transient Ischemic Attack; Atherosclerosis; Stenosis; Stents
Keywords: Stroke; Transietn Ischemic Attack; Stents; Stenosis
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Atherosclerosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Stent implantation (Wingspan, Coroflex, and TiTAN2)
- 2 (Active Comparator)
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Device: Stent implantation (Wingspan, Coroflex, and TiTAN2) — Stent Implantation:
  Wingspan intracranial stent with Gateway PTA balloon Catheter; Coroflex&reg - balloon expandable stent system and Coroflex Blue - Coronary Stent System; TiTAN2 Bio-active coating stent
  Standard Medical Management:including antiplatelet agents(Aspirin 75~150mg/day or Clopidogrel 75mg/day),statins(Atorvastatin 20mg/day or Simvastatin 20mg/day),risk factor lowering agents (antihypertension agents:Amlodipine 5mg/day or Benazepril 10mg/day or Valsartan 80mg/day or Nifedipine 30mg/day or Indapamide 2.5mg/day,antidiabetic agents: Metformin 0.5 tid or Glipizide 5mg tid or Acarbose 50mg tid )if necessary,interactive education program (Online medical education program, health behavior guide) .
  Arms: 1
  Arms: 1
Drug: Standard medical treatment — Standard Medical Management:including antiplatelet agents(Aspirin 75~150mg/day or Clopidogrel 75mg/day),statins(Atorvastatin 20mg/day or Simvastatin 20mg/day),risk factor lowering agents (antihypertension agents:Amlodipine 5mg/day or Benazepril 10mg/day or Valsartan 80mg/day or Nifedipine 30mg/day or Indapamide 2.5mg/day,antidiabetic agents: Metformin 0.5 tid or Glipizide 5mg tid or Acarbose 50mg tid )if necessary,interactive education program (Online medical education program, health behavior guide)
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of stent implantation in patients with symptomatic extra- and intracranial artery stenosis and to determine its role in secondary prevention of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between above 40 year-old and 75 year-old.
2. Ischemic stroke related to extra- and intracranial atherosclerosis stenosis, transient ischemic attack (TIA ), onset time within 90 days
3. Implantation of stent should be at least 1 week after stroke onset, and patient's medical condition stable, no time limit for TIA,
4. Stenosed ICA or MCA or BA or VA is the candidate arteries for stent implantation.
5. Degree of stenosis of target artery ranges between 51%-99%
6. Modified Rankin score≤3 or NIHSS Score ≤4
7. Informed consent is obtained.

Exclusion Criteria:

Patients will be excluded from entry if any of the criteria listed below are met:

1. Target stenosis artery is not suitable for stent implantation after evaluation.
2. Previous carotid endarterectomy or carotid artery stent ,or intracranial artery stent implantation.
3. Ischemic stroke is caused by conditions other than atherosclerosis .
4. Documented non-atherosclerosis angiopathy.
5. Clinically unstable at the time of enrollment,
6. Conditions which may lead to cardiogenic embolism : arterial fibrillation，left ventricular thrombi,Myocardiac infarction within 6 weeks,etc.
7. Severe hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg)
8. Severe co-morbid or unstable medical condition, ie，severe heart failure, pulmonary failure or renal failure, liver dysfunction (serum liver enzyme twice or more than normal level),malignancy with likelihood of death within the next 2 years
9. Significant memory or behavioral disorder, ie, Alzheimer disease, etc.daily care needed.
10. Concurrent participation in another clinical trial
11. Unable to return follow up
12. History of hemorrhagic disease(ie, intracranial hemorrhage, Idiopathic Thrombocytopenic Purpura,etc ) or bleeding tendency conditions.
13. Intracranial arteriovenous malformation or aneurysm.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke in the supply area of stent implantation artery | 30 days and 1 year after the procedure

SECONDARY OUTCOMES:
Hemorrhagic stroke | 30 days and 1 year after the procedure
Ischemic stroke in the supply area of non-stent implantation artery | 30 days and 1 year after the procedure
Acute coronary syndrome | 30 days and 1 year after the procedure
All-cause death | 30 days and 1 year after the procedure
Transient ischemic attack | 30 days and 1 year after the procedure
Degree of re-stenosis of the stent implantation artery | 30 days and 1 year after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Liying Cui, Principal Investigator — Peking Union Medical College Hospital
Locations (10):
- China (10):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital, Chongqing, Chongqing Municipality
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Jilin University, Changchun, Jilin
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Center of Medical Sciences, Chengdu, Sichuan
  - The General Hospital Under Tianjin Medical Sciences University, Tianjin, Tianjin Municipality